CLINICAL TRIAL: NCT03143569
Title: Ventricular Assist Device Anti-Factor Xa (VAD ANTIX) Monitoring Study: a Prospective Randomized Feasibility Trial
Acronym: VAD-ANTIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Thomas Graetz, Assoc Prof of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201701126
Record Dates: First submitted 2017-04-20; First posted 2017-05-08 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Left Sided Heart Failure; Left Ventricular Assist Device; Anticoagulant Therapy; Gastro Intestinal Bleeding; Thrombosis, LVAD; Anti-factor Xa; aPTT; Heparin
MeSH Terms: conditions — Heart Failure; Gastrointestinal Hemorrhage; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- aPTT nomogram (Active Comparator): aPTT guided heparin management
  Interventions: Device: aPTT guided heparin management; Device: Anti-factor Xa guided heparin management
- Anti-factor Xa nomogram (Experimental): Anti-factor Xa guided heparin management
  Interventions: Device: aPTT guided heparin management; Device: Anti-factor Xa guided heparin management

INTERVENTIONS:
Device: aPTT guided heparin management — post-surgical implantation anti-coagulation therapy to prevent clotting in ventricular assist device.
Device: Anti-factor Xa guided heparin management — post-surgical implantation anti-coagulation therapy to prevent clotting in ventricular assist device

SUMMARY:
This study evaluates two different methods for monitoring a patient's anti-clotting [heparin] therapy after they receive a heart pump implant [left ventricular assist device -LVAD]. One method tests for how long it takes the patient's blood to clot and uses that to determine if they are on the right dose of heparin. The other method uses a more direct measure of how much heparin is in the blood. The hypothesis is that the method that more directly measures how much heparin is in the patient's blood will provide better medical results for the patient's care after they have the heart pump implant. To that end, the investigators are conducting this feasibility trial to establish the logistics associated with the implementation of these heparin monitoring approaches.

DETAILED DESCRIPTION:
Heart failure is a medical condition that is on the rise in the US and is associated with an enormous cost of $30 billion in healthcare expenses. People with heart failure may be treated with an LVAD that is connected to their heart and helps it pump the blood from the left side of the heart into the blood vessels that delivers blood to the body. These devices can be used to treat heart failure for the long term or they can be used while a patient waits for a heart transplant. In either case, the use of these devices is increasing.

One of the primary risks associated with LVADs are those related to blood clotting. Maintenance of the LVAD depends on preventing blood clots especially right after the surgery that puts them in place. This requires putting patients with LVADs on blood thinners and then monitoring the blood thinner levels carefully so that they don't have problems with bleeding too easily or, on the other hand, forming blood clots if they aren't on the right dose of blood thinners. Excessive bleeding - called hemorrhaging - is the more common problem after surgery and half of all patients that receive an LVAD will require a blood transfusion within the first 30 days after they receive the device. A laboratory test that measures how quickly blood clots is used to determine if the patient has the right amount of blood thinners. The current standard test is called "activated partial thromboplastin time [aPTT]." There are problems with the reliability of this test because it reacts with other elements in the blood. Alternately, there is a test that more directly measures the amount of heparin blood thinner rather than coagulation time and may be more reliable than aPTT called anti-factor Xa [anti-Xa].

The investigators have developed process diagrams that show steps for making decisions [called nomograms] that tell a nurse or doctor how to manage the heparin levels using test results from the aPTT test or the anti-Xa test; however, both tests will be performed at each decision time point, but the care team will only be told the results from the testing to which their patient is assigned.

The purpose of this feasibility study is to establish feasibility of using the two nomograms to determine which provides the optimal clinical information for improving patients' outcomes that have had LVADs placed.

Potential subjects will be recruited prior to their surgery and may decline to participate anytime before or after the surgery takes place. Subjects will be randomized to the aPTT nomogram or the anti-Xa nomogram. If they withdraw consent, they will receive the aPTT standard of care monitoring. The study procedures are performed by the clinical care team. Clinicians will be trained to use the nomograms.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Implantation with HeartMate II® or HeartWare®, LVAD at Barnes Jewish Hospital

Exclusion Criteria:

1. Unable to receive heparin-based therapy
2. Hypercoagulable disorders [factor V Leiden, Antithrombin deficiency, Protein C deficiency, Antiphospholipid antibodies or other thrombophilia]
3. Incarceration
4. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Graetz, MD, Principal Investigator — Dept of Anesthesiology, Washington University STL SOM
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: 10 patients, that met all inclusion and exclusion criteria, were enrolled in each arm
Groups:
- Total: Total of all reporting groups
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.3) | 50.5 (13.4) | 51.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
INTERMACS Profile score less than 4 [Count of Participants; unit: Participants] — INTERMACS(R) (Interagency Registry of Mechanically Assisted Circulatory Support) patient profile at the time of implant is a general description of patients receiving LVADs. INTERMACS(R) profile 1 is in Critical cardiogenic shock. INTERMACS(R) profile 2 is in Progressive decline. INTERMACS(R) profile 3 is Stable but inotrope dependent. INTERMACS(R) profile 4 is Resting symptoms. INTERMACS(R) profile 5 is Exertion intolerant. INTERMACS(R) profile 6 is Exertion limited. INTERMACS(R) profile 7 is Advanced NYHA Class 3. The lower the INTERMACS(R) profile, the more severe their heart failure.
  Participants | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Nomogram Feasibility
Description: Questionnaires evaluating pragmatic application of nomograms. Question 1: The current heparin nomogram using (aPTT or anti-Xa depending on group) monitoring is easy to follow.
Time Frame: 14 days of heparin therapy
Measure: Number; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (Surveys) | 136 | 112
Surveys
  Surveys Completed | 136 | 112
  Affirmative Responses | 136 | 111
Statistical Analysis 1: Comparison: aPTT Nomogram vs Anti-factor Xa Nomogram; Test type: Other; p = .45, Fisher Exact

2. Primary Outcome: Nomogram Feasibility
Description: Questionnaires evaluating pragmatic application of nomograms. Question 2: Overall, I am satisfied with the utilization and implementation of the heparin monitoring nomogram.
Time Frame: 14 days of heparin therapy
Population: Collected Survey responses from bedside nurses. All surveys were collected as intended.
Measure: Number; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (Surveys) | 136 | 112
Surveys
  Surveys Completed | 136 | 112
  Affirmative Responses | 136 | 112
Statistical Analysis 1: Comparison: aPTT Nomogram vs Anti-factor Xa Nomogram; Test type: Other; p = 1.0, Fisher Exact

3. Primary Outcome: Nomogram Feasibility
Description: Questionnaires evaluating pragmatic application of nomograms. Question 3: Overall, I feel that this dosing nomogram is feasible.
Time Frame: 14 days of heparin therapy
Population: Collected Survey responses from bedside nurses. All surveys were collected as intended.
Measure: Number; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (Surveys) | 136 | 112
Surveys
  Surveys Completed | 136 | 112
  Affirmative Responses | 135 | 112
Statistical Analysis 1: Comparison: aPTT Nomogram vs Anti-factor Xa Nomogram; Test type: Other; p = 1.0, Fisher Exact

4. Primary Outcome: Nomogram Feasibility
Description: Questionnaires evaluating pragmatic application of nomograms. Question 4: When my patient is on the heparin nomogram, I follow the dosing and monitoring instructions exactly.
Time Frame: 14 days of heparin therapy
Measure: Number; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (Surveys) | 136 | 112
Surveys
  Surveys Completed | 136 | 112
  Affirmative Responses | 136 | 112
Statistical Analysis 1: Comparison: aPTT Nomogram vs Anti-factor Xa Nomogram; Test type: Other; p = 1.0, Fisher Exact

5. Primary Outcome: Nomogram Feasibility
Description: Questionnaires evaluating pragmatic application of nomograms. Question 5: I often had to seek clarification from a coworker, pharmacist, NP, or MD regarding the nomogram instructions.
Time Frame: 14 days of heparin therapy
Measure: Number; unit: Surveys
Units Other Than Participants: Surveys
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (Surveys) | 136 | 112
Surveys
  Surveys Completed | 136 | 112
  Affirmative Responses | 45 | 22
Statistical Analysis 1: Comparison: aPTT Nomogram vs Anti-factor Xa Nomogram; Test type: Other; p = .018, Chi-squared

6. Primary Outcome: Success of Nomogram
Description: Amount of time sustained in therapeutic anticoagulation range
Time Frame: 14 days of heparin therapy
Population: Each group received heparin anticoagulation and had heparin administration guided by a nomogram based on one of two different laboratory assays, aPTT or anti-Xa.
Measure: Median (Inter-Quartile Range); unit: % of time patients test was therapeutic
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
% of time patients test was therapeutic | 39.8 [33.3 to 53.3] | 55.8 [50.0 to 63.5]

7. Secondary Outcome: Nomogram Concordance
Description: Compare heparin dosing success between aPTT and anti-factor Xa nomograms. If aPTT was within therapeutic range of nomogram AND anti-factor Xa was within range in therapeutic nomogram, then paired values were deemed "concordent". Similiarly if both aPTT AND anti-factor Xa were above therapeutic range OR both below therapeutic range, then paired valued were deemed "concordent". Otherwise values deemd "discordant"
Time Frame: 14 days of heparin therapy
Population: paired aPTT samples compared with antiXa samples
Measure: Count of Units; unit: tests
Units Other Than Participants: tests
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
Number analyzed (tests) | 416 | 416
tests
  subtherapeutic | 242 | 166
  therapeutic | 138 | 223
  supratherapeutic | 36 | 27

8. Secondary Outcome: Dosing Changes
Description: Number of dosing changes during heparin therapy until first therapeutic
Time Frame: 14 days of heparin therapy
Measure: Median (Inter-Quartile Range); unit: dosing changes
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
dosing changes | 4.0 [1.0 to 7.0] | 3.0 [1.0 to 4.0]

9. Secondary Outcome: Time to Therapeutic Dose
Description: Amount of time needed to achieve therapeutic dose from heparin initiation
Time Frame: 14 days of heparin therapy
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
Number analyzed (Participants) | 10 | 10
hours | 48.0 [12.0 to 60.0] | 33.0 [6.0 to 48.0]

ADVERSE EVENTS:
Time Frame: Collected during 14 day study duration.
Arm/Group | aPTT Nomogram | Anti-factor Xa Nomogram
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 3/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aPTT Nomogram (N=10) | Anti-factor Xa Nomogram (N=10)
Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 3 (3) — Thrombotic events
Bleeding Complication (Blood and lymphatic system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT03143569/Prot_SAP_000.pdf